CLINICAL TRIAL: NCT03679780
Title: The Effect of Endothelin and L-Arginine on Racial Differences in Vasoconstriction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Matthew Brothers, Associate Professor, The University of Texas at Arlington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-0648
Record Dates: First submitted 2018-09-17; First posted 2018-09-20 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; Vasoconstriction
Keywords: Racial Differences; Oxidative Stress
MeSH Terms: conditions — Cardiovascular Diseases | interventions — BQ 788; cyclo(Trp-Asp-Pro-Val-Leu); Arginine; NG-Nitroarginine Methyl Ester; Nitroprusside; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Each subject has one control site and three experimental sites concurrently tested within the same study using intradermal microdialysis on the dorsal forearm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator): This site will serve as the control site and will receive lactated Ringer's (saline solution) (2 µl/min) throughout the entire duration of the protocol. This site will additionally receive 20mM L-NAME and 28mM SNP to inhibit nitric oxide (NO) production and elicit vasodilation, respectively, to assess NO contribution and maximal vasodilation.
  Interventions: Drug: NG Nitro L Arginine Methyl Ester; Drug: Sodium Nitroprusside; Drug: Lactated Ringer's
- Inhibitor of Endothelin Type B Receptor (Experimental): This site will receive 300 nM BQ-788, an inhibitor of the endothelin type B receptors. This site will additionally receive 20mM L-NAME and 28mM SNP to inhibit nitric oxide (NO) production and elicit vasodilation, respectively, to assess NO contribution and maximal vasodilation.
  Interventions: Drug: BQ-788; Drug: NG Nitro L Arginine Methyl Ester; Drug: Sodium Nitroprusside
- Inhibition of Endothelin Type A Receptor (Experimental): This site will receive 500 nM aBQ-123, an inhibitor of endothelin type A receptors. This site will additionally receive 20mM L-NAME and 28mM SNP to inhibit nitric oxide (NO) production and elicit vasodilation, respectively, to assess NO contribution and maximal vasodilation.
  Interventions: Drug: BQ-123; Drug: NG Nitro L Arginine Methyl Ester; Drug: Sodium Nitroprusside
- L-Arginine (Experimental): This site will receive 10 mM L-Arginine to supplement the substrate for endothelial nitric oxide synthase. This site will additionally receive 20mM L-NAME and 28mM SNP to inhibit nitric oxide (NO) production and elicit vasodilation, respectively, to assess NO contribution and maximal vasodilation.
  Interventions: Drug: L-Arginine; Drug: NG Nitro L Arginine Methyl Ester; Drug: Sodium Nitroprusside

INTERVENTIONS:
Drug: BQ-788 — This intervention is aimed at blocking endothelin type B receptors to assess racial differences during vasoconstriction. The infusion rate will be 2 µl/min
  Arms: Inhibitor of Endothelin Type B Receptor
Drug: BQ-123 — This intervention is aimed at blocking endothelin type A receptors to assess racial differences during vasoconstriction. The infusion rate will be 2 µl/min
  Arms: Inhibition of Endothelin Type A Receptor
Drug: L-Arginine — A substrate that is administered to increase endogenous nitric oxide production. The infusion rate will be 2 µl/min
  Arms: L-Arginine
Drug: NG Nitro L Arginine Methyl Ester — L-Name is a NOS inhibitor that is administered to each site to allow for the quantification of NO contribution to vasodilation. The infusion rate will be 2 µl/min
  Other Names: L-Name
Drug: Sodium Nitroprusside — SNP will be perfused through each site to induce maximal vasodilation. The infusion rate will be 2 µl/min
  Other Names: SNP
Drug: Lactated Ringer's — Lactated Ringer will serve as the control site. The infusion rate will be 2 µl/min
  Arms: Control

SUMMARY:
The goal of the study is to examine the possible mechanisms of impaired cutaneous microvascular function through local heating along with administration of vasoconstrictors.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) afflicts nearly one-third of the adult population with all races and ethnicities represented in CVD prevalence. Unfortunately, a disparity exists such that the black population (BL) is disproportionately affected compared to other groups, including the white population (WH). While the underlying cause of this disparity is multifactorial, vascular dysfunction (i.e., impaired vasodilation and/or augmented vasoconstriction) is a key contributor. Across a series of studies conducted in our laboratory we have consistently observed impaired microvascular function in the small blood vessels in the skin (the cutaneous microvasculature) in AA relative to age, sex, and body mass index Caucasian Americans (CA). From a research design perspective this offers the opportunity to conduct minimally invasive studies while investigating research questions in a systematic and mechanistic manner. Furthermore, the cutaneous circulation is recognized as surrogate vascular bed for assessment of mechanisms underlying systemic vascular disease and microvascular dysfunction is emerging as a critical step in the artherosclerotic process and a variety of conditions including hypertension, exercise intolerance, and insulin resistance. And, impaired cutaneous microvascular function mirrors impaired responses in other vascular beds. A primary advantage to utilizing the cutaneous circulation is that it provides an accessible vascular bed through which processes of endothelial function can be investigated, with virtually no risk, through thermal stimuli and local intra-dermal drug infusions.

In terms of the AA population our group and others have documented that impaired vascular function and elevated disease risk is related, in part, to reductions in bioavailability of the potent vasodilator Nitric oxide (NO). While, this has become fairly common knowledge what remains less well defined is the mechanisms of this reduced NO bioavailability. We have recently identified a role for oxidative stress in this process. However, oxidative stress is a complex process and likely does not explain all of the observed impairment. 2 other possibilities that are attractive candidate targets for mechanistic studies are the endothelin pathway as well as bioavailability of L-Arginine. Endothelin is a hormone that has been implicated in many populations with elevated CVD risk as it is a potent vasoconstrictor which also can reduce NO bioavailability. Interestingly, there are reports of elevated endothelin circulating concentration and/or increased sensitivity and thus vasoconstriction to endothelin in AA. L-Arginine is a naturally occurring amino acid that is required for the full endogenous production of NO. In other words reduced L-Arginine bioavailability is present in many disease conditions and contributes to vascular dysfunction. In regards to AA it is reported that they have reduced natural production of L-arginine and also respond more positively to intra coronary infusion of L-arginine relative to other populations. However, to our knowledge the role of the endothelin system as well as L-arginine in microvascular dysfunction in AA has never been investigated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (ages 18-35, both genders) will be recruited from the greater Arlington area to participate in the study.
* Must self-report both parents as either African American or Caucasian American.

Exclusion Criteria:

* Individuals who have donated more than 550 ml of blood within the past 8 weeks will not have blood drawn from them in this protocol. However, if they remain interested in the study, and otherwise meet the inclusion criteria, than we may still opt to proceed with data collection.
* Individuals with cardiovascular, neurological, and/or metabolic illnesses will be excluded from participating as well as individuals with a history of various diseases of the microvasculature including Reynaud's disease, cold-induced urticaria, cryoglobulinemia, etc.
* Subjects currently taking any prescription medications and individuals with a body mass index about 30 kg/m2) will be excluded.
* Pregnant subjects and children (i.e. younger than 18) will not be recruited for the study. Eligible females will be scheduled for days 2-7 of their menstrual cycle to account for hormonal effects on blood flow. A regular menstrual cycle is required to identify and schedule the study for the low hormone period, therefore females who lack a regular cycle will be excluded from the study. Females currently taking birth control are eligible, as long as they can be scheduled during a low-hormone "placebo" week. If their hormone do not contain a placebo week than these individuals will not be eligible for data collection. Females who are breast-feeding will also be eligible as there are no systemic or lasting effects of the proposed vasoactive agents.
* Given that smoking can affect the peripheral vasculature, current smokers and individuals who regularly smoked (>1 pack per two weeks) within the prior 2 years will be excluded

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Vasodilatory Response to Endothelin Receptor-A/B Blockers and L-Arginine following local heating as assessed by Intradermal Microdialysis and Laser Doppler Fluxmetry | Through study completion, an average of 1 Year
  Determine to what extent overactivation of Endothelin Receptor Type A/B or L-Arginine deficiencies have on vasodilatory capacity by delivering specific Endothelin receptor agonists or supplemental L-Arginine via intradermal microdialysis. Vasodilation will be elicited by local heating and changes in skin blood flux will be assessed via laser Doppler fluxmetry. All changes in skin blood flux will be normalized and reported as a percentage of maximal flux.

CONTACTS AND LOCATIONS:
Locations (1):
- Science and Engineering Research and Innovation Building, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No